CLINICAL TRIAL: NCT04206345
Title: Acute Effects of Exercises Combined With Blood Flow Restriction on Strength, Proprioception and Functional Motor Performance in Healthy Individuals
Brief Title: Acute Effects of Exercises Combined With Blood Flow Restriction in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gonca Şahiner Pıçak, reaserch assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/18-25
Record Dates: First submitted 2019-11-20; First posted 2019-12-20 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Healthy Individuals
Keywords: blood flow restriction; acute
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood Flow Restriction Group (Experimental): Elbow bending exercises with resistance exercise band (%20 of 1 maximum repetition) for one session. Blood flow restriction band will be placed during exercise session. The first set of exercises will be 30 repetitions then 3 sets of 15 repetitions. Totally 75 repetitions will be performed. 30 seconds rest interval between sets will be given.
  Interventions: Other: exercise with blood flow restriction
- Exercise Group (Experimental): Elbow bending exercises with resistance exercise band (%70 of 1 maximum repetition) will be performed for one session.
  Interventions: Other: exercise
- Control Group (No Intervention): 10 minutes resting period will be given between evaluation.

INTERVENTIONS:
Other: exercise with blood flow restriction — Elbow bending exercises with blood flow restriction will be performed to the exercise group.
  Arms: Blood Flow Restriction Group
Other: exercise — Elbow bending exercises
  Arms: Exercise Group

SUMMARY:
Purpose of the study is; to investigate the acute effects of exercises combined with blood flow restriction on strength, proprioception and functional motor performance in healthy individuals. The investigators hypothesized that blood flow restriction exercises has a positive effect on strength, proprioception and functional motor performance.

DETAILED DESCRIPTION:
60 healthy individuals will randomized into 3 groups of 20 people each. Participants will be held in a familiarization session before 3-4 days the actual evaluation. Elbow bending exercises with blood flow restriction will be performed to the blood flow restriction (BFR) group, elbow bending exercises without blood flow restriction will be performed to the exercise group and control group will not receive any interventions. Participants will be evaluated before and after the exercise session. Control group is going to rest for 10 minutes before the second evaluation. Evaluation protocol includes; muscle strength measurement with digital hand dynamometer, shoulder and elbow proprioception evaluation with inclinometer, Upper Extremity Closed Kinetic Chain Stabilization Test, Functional Throwing Performance Index and Modified Pull-Up Test.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Do not smoke
* Having full range of motion in neck, shoulder, and elbow
* Body mass index (BMI)˂30 kg/m2
* Able to complete the entire study procedure

Exclusion Criteria:

* Having fracture and surgical history for the upper extremity, cervical or thoracic area
* Having any systemic musculoskeletal disease
* Having neck and upper extremity pain
* Having a diagnosis of scoliosis and chest deformity
* Regularly playing sports with overhead activities (tennis, volleyball, handball, etc.)
* Have been exercising regularly for the last 6 months
* A history of anemia
* A history of cerebrovascular disease or myocardial infarction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Strength | baseline measurements and after 10 minutes of one exercise session
  Change of biceps muscle strength(in kg, with hand held dynamometer)

SECONDARY OUTCOMES:
Shoulder proprioception | baseline measurements and after 10 minutes of one exercise session
  Change of shoulder proprioception for 100 abduction (with bubble inclinometer)
Elbow proprioception | baseline measurements and after 10 minutes of one exercise session
  change of elbow proprioception for three degrees: 45, 60 and 75 (with digital inclinometer)
Modified Pull-Up Test | baseline measurements and after 10 minutes of one exercise session
  Number of pull-ups will be recorded
Upper Extremity Closed Kinetic Chain Stabilization Test | baseline measurements and after 10 minutes of one exercise session
  This test will be occurred in plank position. Participant will touch with one hand to other while maintaining the position. Number of touch will be recorded.
Functional Throwing Performance Index | baseline measurements and after 10 minutes of one exercise session
  Participants will throw a ball to shot a frame on a wall. Number of correct shots will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Yesilyaprak, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, Select State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No